CLINICAL TRIAL: NCT05893485
Title: Physiological and Psychological Effects of Music Therapy in the Pregnant Woman and Fetus, WOMB (Women on Musical Bedrest)
Brief Title: Physiological and Psychological Effects of Music Therapy in the Pregnant Woman and Fetus
Acronym: WOMB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christina Chianis Reed (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor-Investigator, Christina Chianis Reed, Assistant Professor of OB/GYN, Dir of Ops Placenta Accreta Care Team, and Dir of Clinical Research, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-52059
Record Dates: First submitted 2023-01-17; First posted 2023-06-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Music Therapy; Preterm Premature Rupture of Membrane (PPROM)
Keywords: Music therapy; Antepartum; Preterm Premature Rupture of Membranes (PPROM); Fetus; Woman; Post Traumatic Stress Disorder; Postpartum Depression; Anxiety; Stress
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes; Stress Disorders, Post-Traumatic; Depression, Postpartum; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): No Music Therapy
- Music Therapy Intervention (Active Comparator): Four music therapy sessions provided prior to delivery.
  Interventions: Behavioral: Music Therapy Intervention

INTERVENTIONS:
Behavioral: Music Therapy Intervention — Music Therapy Sessions. There will be 4 scheduled music therapy sessions, and a postpartum follow up.
  Arms: Music Therapy Intervention

SUMMARY:
To evaluate the effects of music therapy in the care of antepartum mothers admitted for long-term hospitalization due to the high-risk status of their pregnancy. The investigators speculate that mothers who receive music therapy will be more successful in forming positive coping habits, bonding with their infant, and increasing the length of incubation during their pregnancy.

Furthermore, there is no research that correlates music therapy applied to stress reduction, increased coping, and increased caregiver-infant bonding prior to birth within one protocol. However, there is a significant amount of research supporting music therapy efficacy with neonatal intensive care unit infants and caregiver bonding post-partum as well as improved physiological signs of stress in infants in the post-partum period.

DETAILED DESCRIPTION:
The investigators will identify and screen patients who are admitted to the Texas Children's Pavilion for Women and Houston Methodist Willowbrook with a clinical diagnosis of threatened preterm birth caused by preterm premature rupture of membranes (PPROM), between a gestational age of 24 and 36 weeks. The investigators will approach the patients to discuss this study and if they are interested in participating, the investigators will provide the informed consent form for their signature. After that, the investigators will start collecting data, such as basic demographic information and the Edinburgh Postnatal Depression Scoring scale (EDPS) scores that are clinically taken before and after the PPROM diagnosis.

Inclusion Criteria:

1. Pregnant women between 18 and 64 years of age.
2. Singleton pregnancy.
3. Hospital admission due to a high risk of premature delivery.
4. Confirmed diagnosis of preterm premature rupture of membranes.
5. Length of stay in the hospital for 48 hours or more and stable for 48 hours or more.
6. Patients willing to listen to music.
7. Patients willing to participate throughout all the music therapy sessions and the postpartum follow-up visit.

Exclusion Criteria:

1. Hospital length of stay of less than 48 hours.
2. Non-singleton pregnancy.
3. Gravidae with severe medical and or surgical complications during their hospital admission that prevents them from participating in Music Therapy sessions.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women between 18 and 64 years of age.
2. Singleton pregnancy.
3. Hospital admission due to a high risk of premature delivery.
4. Confirmed diagnosis of preterm premature rupture of membranes.
5. Length of stay in the hospital for 48 hours or more and stable for 48 hours or more.
6. Patients willing to listen to music.
7. Patients willing to participate throughout all the music therapy sessions and the postpartum follow-up visit.

Exclusion Criteria:

1. Hospital length of stay of less than 48 hours.
2. Non-singleton pregnancy Gravidae with severe medical and or surgical complications during their hospital admission that prevents them from participating in Music Therapy sessions.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Measure the length of time from when the membranes prematurely rupture to delivery | 30 days
  Time will be measured in hours from when the membranes prematurely rupture between 24 and 34 weeks of gestational age. The time will be compared to those who do not receive music therapy. The shorter the time interval means worse outcomes.

SECONDARY OUTCOMES:
Change in anxiety levels in relation to the length of hospital stay | 30 days
  Determine if there is a relationship between anxiety levels and hospital length of stay. The hospital length of stay is measured by hours spent in-patient at the hospital. Anxiety levels will be assessed using the Visual Analogue Scale for Anxiety. The Visual Analogue Scale for Anxiety is a 10 centimeter line with the minimum score of "not at all anxious" to the left and the maximum score of "very anxious" to the right. The more anxious a person is they put a mark on closer to "very anxious" which is the worse outcome.
Music therapy in relation to maternal tachycardia due to stress | 30 days
  Determine if music therapy sessions change heart rate on tachycardic women with reported stress.
Edinburgh Postnatal Depression Scale score before and after music therapy | 30 days
  Evaluate the Edinburgh Postnatal Depression Scale scores before and after music therapy. The minimum score is 0 and the maximum score is 30. Possible depression is 10 or greater. Greater the score the worse the outcome. Always look at question number 10 regarding suicidal thoughts.
Visual analogue scale for anxiety before and after music therapy | 30 days
  Correlate the Visual Analogue Scale measuring the state anxiety (VAS-A) scores both antepartum and postpartum in patients who receive music therapy. The Visual Analogue Scale for Anxiety is a 10 centimeter line with the minimum score of "not at all anxious" to the left and the maximum score of "very anxious" to the right. The more anxious a person is they put a mark on closer to "very anxious" which is the worse outcome.
Music therapy in relation to infant bonding | 30 days
  Participants express increased connection/bonding with their infant through a questionnaire given to them at their 6 week postpartum visit. The question has yes or no answers. The participant will choose yes if they feel an increased connection/bonding with their infant and participants will choose no if they do not feel an increased connection/bonding with their infant. The answer choice no is the worse outcome.
Change in the time interval between delivery and newborn receiving their mother's breastmilk | 30 days
  Change in the time interval between delivery and newborn receiving their mother's breastmilk normalized to gestational age at delivery.
Change in blood pressure before and after music therapy | 30 days
  Measure blood pressure at pre-determined times before and after music therapy. Higher blood pressure is a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Reed, WHNP-BC, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Pavilion for Women, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Corey K, Fallek R, Benattar M. Bedside Music Therapy for Women during Antepartum and Postpartum Hospitalization. MCN Am J Matern Child Nurs. 2019 Sep/Oct;44(5):277-283. doi: 10.1097/NMC.0000000000000557. PMID 31274510
- [Background] Teckenberg-Jansson P, Turunen S, Pölkki T, et al. Effects of live music therapy on heart rate variability and self-reported stress and anxiety among hospitalized pregnant women: A randomized controlled trial. Nordic Journal of Music Therapy. 2019; 28(1): 7-26.
- [Background] Yang M, Li L, Zhu H, Alexander IM, Liu S, Zhou W, Ren X. Music therapy to relieve anxiety in pregnant women on bedrest: a randomized, controlled trial. MCN Am J Matern Child Nurs. 2009 Sep-Oct;34(5):316-23. doi: 10.1097/01.NMC.0000360425.52228.95. PMID 19713801